CLINICAL TRIAL: NCT00841022
Title: Effects of Comics on Anaesthesia's Anxiety in Paediatrics: A Randomized Controlled Trial
Brief Title: Information and Anaesthesia in Paediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008.518
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-10

CONDITIONS: Anxiety
Keywords: anxiety; anaesthesia; child; RCT; Elective surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Information of children with comic leaflet
  Interventions: Other: Information with comics
- 2 (No Intervention)

INTERVENTIONS:
Other: Information with comics — Information of children with comic leaflet
  Arms: 1

SUMMARY:
This study aims to investigate whether detailed and illustrated information (comics) about anaesthesia reduce preoperative anxiety in children being subjects to craniotomy.

Children scheduled for craniotomy are randomized to groups receiving a comic leaflet explaining the course of anaesthesia before preanaesthesia visit or no intervention.

Preoperative anxiety is assessed with anxiety scale STAIC for the two groups of participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children between 6 to 16 years and 11 month old.
* Children scheduled to have a craniotomy or orthopaedic surgery (multi-level surgery, spinal decompression, osteosarcoma resection, column surgery , fibroid curettage, Nuss bar procedure, hip varus surgery) or visceral and urologic surgery (intestinal continuity restoration, hypospadias surgery, bladder malformation, sarcoma).
* Children with a high, normal or light level of verbal comprehension (normal academic level or less than two repeating).
* Children coming with their parents.

Exclusion Criteria:

* Previous surgery.
* Unwillingness to participate (parents or child)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2009-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Level of anxiety scale (STAIC-S) | before preanaesthesia consultation and after preanaesthesia consultation

SECONDARY OUTCOMES:
Level of verbal comprehension : WISC 4 (similitude, vocabulary and comprehension) | before preanaesthesia consultation
Level of anxiety scale (STAIC-T) | Before preanaesthesia consultation

CONTACTS AND LOCATIONS:
Overall Officials: Edmundo PEREIRA DE SOUZA NETO, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Kassai B, Rabilloud M, Dantony E, Grousson S, Revol O, Malik S, Ginhoux T, Touil N, Chassard D, Pereira de Souza Neto E. Introduction of a paediatric anaesthesia comic information leaflet reduced preoperative anxiety in children. Br J Anaesth. 2016 Jul;117(1):95-102. doi: 10.1093/bja/aew154. PMID 27317708